CLINICAL TRIAL: NCT05159791
Title: New Patient-specific Functional Assessment of the Anomalous Aortic Origin of Coronary Arteries.
Acronym: NECESSARY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Mauro Lo Rito, Pediatric Cardiac Surgeon and Research Associate, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GR-2019-12369116
Record Dates: First submitted 2021-11-16; First posted 2021-12-16 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-03

CONDITIONS: Anomalous Coronary Artery Origin; Anomalous Coronary Artery Arising from the Opposite Sinus; Anomalous Coronary Artery Course; Anomalous Coronary Artery with Aortic Origin and Course Between the Great Arteries; Sudden Cardiac Death; Myocardial Ischemia
Keywords: Fluid mechanics studies of circulation; Fluid mechanics studies of microcirculation; Fluid mechanics studies of transport systems; Biomechanics; Computational fluid dynamics; Hemodynamics; Mathematical modeling; Simulation; Ventricular remodeling; Tissue and organ mechanics; Mechanics of injury; Coronary congenital anomalies; Coronary blood flow assessment; Personalized functional risk assessment; Computaional fluid dynamics; Structural finite element analysis; Integration of multimodal imaging
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Ischemia; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anomalous coronary blood flow (Experimental): Subjects suspected to have AAOCA will be submitted to angiographic coronary CT imaging to confirm the diagnosis. If the diagnosis of AAOCA will be confirmed, subjects will undergo to invasive coronary blood flow evaluation (intervention).
  Interventions: Diagnostic Test: Invasive coronary blood flow assessment and simulations and fluid dynamic patient specific simulation

INTERVENTIONS:
Diagnostic Test: Invasive coronary blood flow assessment and simulations and fluid dynamic patient specific simulation — The coronary blood flow and its distribution between the anomalous and normal artery will be measured by invasive coronary catheterization. Coronary artery flow will be calculated based on intravascular ultrasound (IVUS) and pressure difference measurements. After the IVUS assessment, a pressure transducer (FFR/iFR probe) will be inserted in the coronary artery for pressure measurements. The measurements will be done in the anomalous and normal coronary arteries in each patient to determine coronary flow distribution. Patient's specific heart parameters will be retrieve from CT, MRI and other diagnostic tests and integrated in the simulation module.

SUMMARY:
Anomalous Aortic Origin of the Coronary Arteries (AAOCA) is a rare congenital disease that may cause sudden death in young subjects. Frequently the first and only presentation is with an acute event (such as myocardial infarction or sudden cardiac deaths) during physical effort. Not only symptoms are often absent, but also provocative tests fail to induce ischemia or related signs, showing in most patients negative results. For these limitations, the decision to undergo corrective surgery is based on the morphologic characteristics without the support of a functional evaluation. The study focused on developing a personalized ischemic risk assessment with the aid of fluid dynamic simulations. The simulation system integrate clinical data from different diagnostic sources and integrate them with coronary blood flow evaluation at rest and during simulated physical effort.

DETAILED DESCRIPTION:
Anomalous Aortic Origin of Coronary Arteries (AAOCA) is a congenital condition where one or more coronary vessels originate from an ectopic site within the aorta, such as the opposite or wrong sinus of Valsalva. Its prevalence in the general population, has been estimated between 0.03% and 0.23% depending on the variant evaluated. The anomalous left or right coronary artery, besides its origin, may take 5 different general courses: interarterial, prepulmonic, subpulmonic, retroaortic or retrocardiac. Each of these forms may be subject to cause myocardial ischemia and subsequent sudden death during physical and sport activity.

In most cases, the disease is silent and does not show any symptoms before the sudden cardiac death event (SCD). Only a few AAOCA subjects report symptoms before SCD that usually occurs unexpectedly after a moderate or intense physical activity. It is extremely hard to study the causing factors in a clinical environment due to the stochastic nature of the myocardial ischemic event and the inability to reproduce the exact effort conditions.

Even when a complete assessment is performed, there is no clinical exam that can reproduce sustained exercise conditions responsible for triggering ischemia and SCD. Even if such an exam would exist and provide adequate results, the risk of SCD exceeds the benefits of having a correct diagnosis.

To overcome all the current diagnostic limitations the ideal diagnostic test has to investigate coronary blood supply, myocardial oxygen demand in relation to the physical activity (intensity and duration) required for triggering an ischemic event, without putting the subjects at risk. To date the only possible way to reproduce such conditions is a subject-specific virtual simulation of aortic root and coronary artery integrated with coronary blood flow simulation able to mimic pressure, flow, and oxygen demand characteristics similar to those of intense exercise, in relation to changes that anomalous coronary undergoes under such conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AAOCA of any age will undergo fluid dynamic simulation
* Patients with age > 14 with diagnosis of AAOCA will undergo to invasive coronary flow measurements
* Informed consent

Exclusion Criteria:

* A presence of major associated congenital heart anomalies
* Contraindication to the execution of the diagnostic examination requested such as age < 14 years for invasive coronary flow measurements

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of myocardial ischemia on simulation model | 3 years
  Assess myocardial ischemia in the patient's specific model during simulated effort correlating coronary artery blood supply to myocardial oxygen demand.

SECONDARY OUTCOMES:
Invasive coronary flow distribution assessment | During clinical diagnostic evaluation, average 3 months after
  Evaluation of coronary blood flow (ml/min) in anomalous coronary artery and in normal coronary artery.
Integration of different coronary artery imaging modality | During clinical diagnostic evaluation, average 6 months
  CT 3D reconstruction of aorta and coronary artery with aorta and coronary artery cross-sectional area (mm2); IVUS coronary artery reconstruction cross-sectional area (mm2); coronary blood flow quantification (ml/min)
Computational fluid dynamic simulation | 3 years
  Correlation between at rest estimated coronary blood flow (patient's specific FSI model) and the measured invasive coronary blood flow (FFR and derived measures).
In vitro effort fluid dynamic simulation | 3 years
  FSI model effort will be simulated by increasing heart rate (bpm) and pressure (mmHg) that will determine changes in coronary artery cross-sectional area (mm2). The outcome of the FSI effort simulation will be measured as changes in coronary artery blood flow (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Lo Rito, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceserani V, Lo Rito M, Agnifili ML, Pascaner AF, Rosato A, Anglese S, Deamici M, Negri J, Corrado C, Bedogni F, Secchi F, Lombardi M, Auricchio F, Frigiola A, Conti M. Lumped-parameter model as a non-invasive tool to assess coronary blood flow in AAOCA patients. Sci Rep. 2023 Oct 14;13(1):17448. doi: 10.1038/s41598-023-44568-8. PMID 37838795